CLINICAL TRIAL: NCT06502522
Title: Effects of Whole-body Electrostimulation on Kidney Function and Physical Capacity of Patients With Chronic Kidney Disease: Randomized Clinical Trial
Brief Title: Effects of Whole-body Electrostimulation on Patients With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Leonhardt Ventures LLC (Industry)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WB-EMS-KIDNEY
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Whole-body neuromuscular electrical stimulation will be administered for three times week for eight weeks, totaling 24 sessions.
  Interventions: Other: Whole-body electrical stimulation
- Control group (No Intervention): No intervention will be carried out.

INTERVENTIONS:
Other: Whole-body electrical stimulation — Symmetrical biphasic current, pulse width of 400 μs, frequency of 75 Hz, contraction time of five seconds and rest time of 10 seconds. The intensity will be individually adjusted to the patient's maximum tolerance limit to reach the motor threshold and the volunteer will be instructed to achieve a score of 7 on the modified BORG scale to ensure a moderate-intense effort. The session time will be 16 minutes, resulting in a total of 64 contractions per session. The progression of overload will only occur with an increase in the intensity of all muscle groups during the sessions.
  Concomitantly with the electrical stimuli, the volunteer will perform exercises for the upper, lower limbs and trunk. After performing neuromuscular electrical stimulation, the patient will remain in the supine position to receive sensory stimulation throughout the body. The parameters used will be: frequency of 20 Hz and pulse width of 400 μs for 44 minutes.
  Other Names: Whole-body electrical muscle stimulation; Whole-body neuromuscular electrical stimulation; Whole-body electromyostimulation
  Arms: Intervention group

SUMMARY:
Chronic kidney disease (CKD) consists of kidney damage, with consequent progressive and irreversible loss of kidney function. In the early stages of the disease, a reduction in circulating levels of the α-klotho protein is already observed, which is related to worsening renal function. Therapeutic strategies that increase serum levels of α-klotho may be of great value in the treatment of CKD. Electrical stimulation contributes to the reduction of reactive oxygen species, DNA damage and improves the effectiveness rate of dialysis, suggesting a systemic effect in patients with terminal CKD. The objective of this study is to evaluate the effects of whole body electrical stimulation on renal function and physical capacity in patients with CKD not dependent on dialysis.

DETAILED DESCRIPTION:
Patients with stage III and IV chronic kidney disease will be randomized into two groups, one group will receive whole-body electrical stimulation and the other group will be a control group (it will only be evaluated and reevaluated at the same times as the intervention group). The intervention group will perform the protocol three times a week, for eight weeks. The following assessments will be conducted pre- and post-intervention: analysis of plasma content of soluble α-Klotho and creatinine to assess renal function; measurement of interleukins and tumor necrosis factor by ELISA to analyze the inflammatory profile; beta-endorphin measurement by ELISA to assess well-being; creatine kinase dosage to assess muscle damage; 10-repetition sit-to-stand test and quadriceps muscle dynamometry to assess lower limb muscle strength; handgrip test with a dynamometer to assess upper limb strength; six-minute walk test to assess functional capacity; application of the EuroQoL-5D questionnaire for quality of life and the Pittsburgh scale to assess sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CKD (≥ 3 months) in stages 3-4 (GFR between 59 and 15 ml/min/1.73m2);
* Age between 18 and 80 years old;
* Functional capacity ≥ 300 meters in the six-minute walk test.

Exclusion Criteria:

* Cognitive dysfunction that prevents assessments from being carried out or inability to understand and sign the informed consent form;
* Intolerance to electrical stimulator and/or changes in skin sensitivity;
* Skin injuries or burns where the electrodes are positioned;
* Patients with stroke sequelae;
* Recent acute myocardial infarction (two months);
* Uncontrolled hypertension (SBP>230 mmHg and DBP>120 mmHg);
* New York Heart Association grade IV heart failure or decompensated;
* Unstable angina or arrhythmia;
* Artificial cardiac pacemaker or implantable cardioverter defibrillator;
* Peripheral vascular changes in the lower limbs such as deep vein thrombosis;
* Disabling osteoarticular or musculoskeletal disease;
* Uncontrolled diabetes (glycemia > 300mg/dL);
* Patients with cancer and/or undergoing oncological treatment;
* Epilepsy;
* Hemophilia;
* Chronic obstructive pulmonary disease;
* Grade II obesity (BMI≥35).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in kidney function | Baseline, after 4 and 8 weeks
  Change in kidney function will be assessed by alpha klotho protein dosage
Change in kidney function | Baseline, after 4 and 8 weeks
  Change in kidney function will be assessed by serum creatinine measurement

SECONDARY OUTCOMES:
Change in inflammatory profile | Baseline, after 4 and 8 weeks
  Change in inflammatory profile will be assessed by measurement of interleukin 6 (IL6)
Change in inflammatory profile | Baseline, after 4 and 8 weeks
  Change in inflammatory profile will be assessed by measurement of interleukin 10 (IL10)
Change in inflammatory profile | Baseline, after 4 and 8 weeks
  Change in inflammatory profile will be assessed by measurement of tumor necrosis factor alpha (TNF-a)
Change in well-being levels | Baseline, after 4 and 8 weeks
  Change in well-being levels will be assessed by serum beta-endorphin dosage
Change in muscle damage levels | Baseline, after 4 and 8 weeks
  Change in muscle damage levels will be assessed by serum creatine kinase (CK) measurement
Change in isometric muscle strength of the quadriceps | Baseline and 8 weeks
  Change in isometric muscle strength of the quadriceps will be assessed by dynamometry
Change in handgrip muscle strength | Baseline and 8 weeks
  Change in handgrip muscle strength will be assessed by dynamometry
Change in lower limb muscle strength | Baseline and 8 weeks
  Change in lower limb muscle strength will be assessed using the 10-repetition sit-and-stand test (10SST)
Change in functional capacity | Baseline and 8 weeks
  Change in functional capacity will be assessed through the distance covered in the six-minute walk test (6MWT)
Change in sleep quality | Baseline and 8 weeks
  Change in sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI).The score ranges from 0 to 21. Lower scores reflect worse sleep quality.
Change in quality of life | Baseline and 8 weeks
  Change in quality of life will be assessed using the EuroQoL-5D (EQ-5D) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jociane Schardong, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre